CLINICAL TRIAL: NCT04488822
Title: Multicenter, Single Arm Study of the Efficacy and Safety of Pexidartinib in Adult Subjects With Tenosynovial Giant Cell Tumor
Brief Title: A Study of the Efficacy and Safety of Pexidartinib in Adult Subjects With TGCT
Acronym: PLX3397
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PL3397-A-A303
Record Dates: First submitted 2020-07-24; First posted 2020-07-28 (Actual); Results first posted 2023-04-27 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Tenosynovial Giant Cell Tumor
Keywords: Tenosynovial Giant Cell Tumor; Pexidartinib; TURALIO™; PLX3397
MeSH Terms: conditions — Giant Cell Tumor of Tendon Sheath | interventions — pexidartinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Pexidartinib (Experimental)
  Interventions: Drug: Pexidartinib

INTERVENTIONS:
Drug: Pexidartinib — 400 mg twice daily for a total daily dose of 800 mg (each capsule contains 200 mg of pexidartinib for oral administration)
  Other Names: TURALIO™; PLX3397

SUMMARY:
This study will assess pexidartinib in adult participants with symptomatic TGCT that is associated with severe morbidity or functional limitations and not amendable to improvement with surgery.

DETAILED DESCRIPTION:
Participants with symptomatic TGCT will be administered pexidartinib 400 mg twice daily continuously with 28-day treatment cycle until criteria for discontinuation are reached. Participants who complete primary endpoint assessments may be eligible to continue receiving pexidartinib until disease progression, unacceptable toxicity, the occurrence of other termination criteria, or withdrawal from the study. Eligible participants' status will be collected every 6 months as a long term follow-up at least 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years (Age ≥ 20 years in Taiwan).
* A diagnosis of TGCT (i) that has been histologically confirmed by a pathologist and (ii) associated with severe morbidity or functional limitations and not amenable to improvement with surgery determined consensually by qualified personnel (eg, 2 surgeons or a multi-disciplinary tumor board).
* Measurable disease as defined by RECIST 1.1 (except that a minimal size of 2 cm is required), assessed from MRI scan by a central radiologist.
* Stable prescription of analgesic regimen during the 2 weeks prior to enrollment.
* Women of childbearing potential must have a negative serum pregnancy test within the 14-day period prior to enrollment (Where demanded by local regulations, this test may be required within 72 hours of enrollment).
* Females of reproductive potential should be advised to use an effective, non-hormonal method of contraception during treatment with pexidartinib and for 1 month after the last dose. Males with female partners of reproductive potential should be advised to use an effective method of contraception during treatment with pexidartinib and for 1 month after the last dose. Female partners of male participants should concurrently use effective contraceptive methods (hormonal or non-hormonal). Women of nonchildbearing potential may be included if they are either surgically sterile or have been postmenopausal for ≥ 1 year. Women who have documentation of at least 12 months of spontaneous amenorrhea and have a follicle stimulating hormone level > 40 mIU/mL will be considered postmenopausal.
* Adequate hematologic, hepatic, and renal function, defined by:

  * Absolute neutrophil count ≥ 1.5 × 10^9/L
  * Hemoglobin > 10 g/dL
  * Platelet count ≥ 100 × 10^9/L
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 1.0 × upper limit of normal (ULN)
  * Total bilirubin and direct bilirubin ≤ 1.0 × ULN
  * Alkaline phosphatase ≤ 1.0 × ULN
  * Creatinine clearance (CLcr) > 15 mL/min
* Willingness and ability to complete the PROMIS Physical Function Scale.
* Willingness and ability to use a diary.
* Willingness and ability to provide written informed consent prior to any study-related procedures and to comply with all study requirements.

Exclusion Criteria:

* Investigational drug/device use within 28 days of enrolment.
* Previous use of pexidartinib or any biologic treatment targeting colony stimulating factor 1 (CSF-1) or the CSF-1 receptor; previous use of oral tyrosine kinase inhibitors are allowed (eg, imatinib or nilotinib).
* Active cancer except for tumor for which a participant is enrolled in the study, (either concurrent or within the last year of starting study drug) that requires therapy (eg, surgical, chemotherapy, or radiation therapy), with the exception of adequately treated basal or squamous cell carcinoma of the skin, melanoma in situ, carcinoma in situ of the cervix or breast, or prostate carcinoma with a prostate-specific antigen value < 0.2 ng/mL.
* Known metastatic TGCT.
* Active or chronic infection with hepatitis C or known positive hepatitis B surface antigen, or known active or chronic infection with human immunodeficiency virus.
* Active liver or biliary tract disease
* Known active tuberculosis.
* Significant concomitant arthropathy in the affected joint, serious illness, uncontrolled infection, or a medical or psychiatric history that, in the Investigator's opinion, would likely interfere with a participant's study participation or the interpretation of his or her results.
* Use of strong Cytochrome P450 (CYP) 3A inducers, including St John's wort, proton pump inhibitors (PPIs), and other products known to cause hepatotoxicity.
* Women who are breastfeeding.
* A screening Fridericia corrected QT interval (QTcF) ≥ 450 ms (men) or ≥ 470 ms (women).
* MRI contraindications.
* History of hypersensitivity to any excipients in the investigational product.
* Inability to swallow capsules.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2021-10-27 (Actual); Study Completion 2026-02-28 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (9):
- China (7):
  - Beijing Ji Shui Tan Hospital, Beijing
  - Peking University Cancer Hospital, Beijing
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Fudan University Shanghai Cancer Center, Shanghai
  - Shanghai General Hospital, Shanghai
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) on completed studies and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Completed studies that has reached a global end or completion with all data set collected and analyzed, and for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Xu H, Wu PK, Ye Z, Fan Z, Li T, Chen TW, Shen J, Yan W, Achiwa I, Yoh K, Kikumori K, Hiruma Y, Greenberg J, Niu X. A Phase 3 Study of the Efficacy and Safety of Pexidartinib in East Asian Patients with Tenosynovial Giant Cell Tumor. Oncol Ther. 2025 Dec;13(4):1025-1039. doi: 10.1007/s40487-025-00365-z. Epub 2025 Aug 21. PMID 40841499

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 40 participants who met all inclusion criteria and no exclusion criteria were enrolled and treated at clinic centers in China and Taiwan. Primary results reported are from baseline up to data cut-off date of 27 Oct 2021. The results presented are based on primary analysis. Data collection is still on-going and additional results will be provided after study completion.
Groups:
- Pexidartinib: Participants who received pexidartinib 400mg twice daily (BID) for a total daily dose of 800 mg (2 capsules in the morning and 2 capsules in the evening).
Period: Overall Study
Arm/Group | Pexidartinib
Started | 40
Completed (Completed = Participants ongoing treatment as of 27 Oct 2021, Not Completed =Participants who discontinued treatment) | 31
Not Completed | 9
Not completed — Adverse Event | 8
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were assessed in the Safety Analysis Set.
Arm/Group | Pexidartinib
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 39
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.9 (12.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 40
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  China | 31
  Taiwan | 9

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) of Pexidartinib Based on RECIST 1.1 of Asian Participants With Symptomatic Tenosynovial Giant Cell Tumor (TGCT) at Week 25
Description: For the assessment of tumor response, participants were classified into the best of the following tumor response categories based on Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) by centrally reviewed MRI scan. Complete response (CR), disappearance of all target lesions and normalization of tumor marker level; partial response (PR), at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters; and overall response rate (ORR), defined as CR+PR, are presented.
Time Frame: At Week 25 postdose
Population: ORR based on RECIST 1.1 was assessed in the Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Pexidartinib
Number analyzed (Participants) | 40
Participants
  CR | 0
  PR | 9
  ORR | 9

2. Secondary Outcome: Overall Response Rate (ORR) of Pexidartinib Based on TVS of Asian Participants With Symptomatic Tenosynovial Giant Cell Tumor (TGCT) at Week 25
Description: For the assessment of tumor response, participants were classified into the best of the following tumor response categories based on Tumor Volume Score (TVS) by centrally reviewed MRI scan. Tumor Volume Score (TVS) is a semi-quantitative MRI scoring system that describes tumor mass and is based on 10% increments of the estimated volume of the maximally distended synovial cavity or tendon sheath involved. A tumor that is equal in volume to that of a maximally distended synovial cavity or tendon sheath was scored 10; a score of 0 indicated no evidence of tumor. Complete response (CR), disappearance of lesion; partial response (PR), at least 50% decrease in volume score relative to baseline; overall response rate (ORR), defined as CR+PR, are presented.
Time Frame: At Week 25 postdose
Population: ORR based on TVS was assessed in the Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Pexidartinib
Number analyzed (Participants) | 40
Participants
  CR | 0
  PR | 19
  ORR | 19

3. Secondary Outcome: Mean Percent Change From Baseline for Range of Motion (ROM) Score in Participants Receiving Pexidartinib
Description: Range of motion (ROM) of the joint was assessed by a qualified, independent, and blinded or third-party assessors at the clinical site. The relative ROM was calculated (expressed in percent) as follows: Relative ROM = 100 x (absolute ROM measured)/(reference ROM standard). The change from baseline in relative ROM at Week 25 was calculated as the difference in relative ROM at Week 25 visit minus relative ROM at Screening visit.
Time Frame: At Week 25 postdose
Population: Mean Percent Change From Baseline for Range of Motion (ROM) was assessed in Full Analysis Set; however, participant assessments falling outside the visit window were excluded from the change from baseline analysis.
Measure: Least Squares Mean (Standard Deviation); unit: Percent Change
Arm/Group | Pexidartinib
Number analyzed (Participants) | 31
Percent Change | 23.05 (3.207)

4. Secondary Outcome: Mean Change From Baseline in the Patient-reported Outcomes Measurement Information System (PROMIS) Physical Function Score in Participants Receiving Pexidartinib
Description: The Patient-reported Outcomes Measurement Information System (PROMIS) physical function scale was used to assess the physical function of the upper and lower limbs. The scale ranges from 1 defined as 'unable to do' or 'cannot do' to 5 defined as 'without any difficulty' or 'not at all', where higher scores represent better outcomes.
Time Frame: At Week 25 postdose
Population: Mean Change From PROMIS was assessed in the Full Analysis Set; however, participant assessments falling outside the visit window were excluded from the change from baseline analysis.
Measure: Least Squares Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pexidartinib
Number analyzed (Participants) | 31
Score on a scale | 0.46 (1.384)

5. Secondary Outcome: Best Overall Response of Pexidartinib Based on RECIST 1.1 and TVS by Centrally Reviewed MRI Scan
Description: Best overall response (CR or PR) of pexidartinib based on RECIST 1.1 and TVS are summarized. Tumor categories for RECIST v1.1 were as follows: complete response (CR), disappearance of all target lesions; partial response (PR), at least a 30% decrease in the sum of diameters of target lesions; stable disease (SD), neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease; progressive disease (PD), at least a 20% increase in the sum of diameters of target lesions; and not evaluable (NE). Tumor categories for TVS were as follows: complete response (CR), disappearance of all target lesions; partial response (PR), at least a 50% decrease in volume score relative to baseline; stable disease (SD), does not meet any of the prior criteria based on score during study; progressive disease (PD), at least a 30% increase in in volume relative to lowest score during the study whether at baseline or some other visit; and not evaluable (NE).
Time Frame: From baseline until disease progression or death (whichever occurs first), up to approximately 29 months
Reporting Status: Not Posted, anticipated posting 2027-02

6. Secondary Outcome: Duration of Response of Pexidartinib Based on RECIST 1.1 and TVS by Centrally Reviewed MRI Scan
Description: Duration of response (DOR) is defined as the date of the first recorded response to the first date of documented disease progression.
Time Frame: Time from the date of first documented response until documented disease progression or death from any cause (whichever occurs first), up to approximately 29 months
Reporting Status: Not Posted, anticipated posting 2027-02

7. Secondary Outcome: Number of Participants Reporting Frequent (≥10%) Treatment-Emergent Adverse Events by Preferred Term
Description: A Treatment-emergent adverse event (TEAE) is defined as an AE that occurs, having been absent before the first dose of study drug, or has worsened in severity or seriousness after the initiating the study drug until post-treatment visit (28 ± 7 days after the last dose of study drug).
Time Frame: Up to approximately 29 months
Reporting Status: Not Posted, anticipated posting 2027-02

8. Secondary Outcome: Area Under the Plasma Concentration Time Curve From Time 0 to 6 Hours AUC(0-6h) in Participants Receiving Pexidartinib
Description: AUC(0-6h) was calculated using standard non-compartmental analysis. AUC(0-6h) for Pexidartinib and primary metabolite, ZAAD-1006a, are presented.
Time Frame: Week 3: Cycle 1 Day 1 at pre-dose, 0.5h, 1h, 2h, 4h, and 6h post-dose (each cycle is 28 days)
Population: AUC(0-6h) was assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Pexidartinib
Number analyzed (Participants) | 7
ng*h/mL
  Pexidartinib | 51500 (28.5)
  ZAAD-1006a | 108000 (52.1)

9. Secondary Outcome: Maximum Plasma Concentration (Cmax) in Participants Receiving Pexidartinib
Description: Cmax was calculated using standard non-compartmental analysis. Cmax for Pexidartinib and primary metabolite, ZAAD-1006a, are presented.
Time Frame: Week 3: Cycle 1 Day 1 at pre-dose, 0.5h, 1h, 2h, 4h, and 6h post-dose (each cycle is 28 days)
Population: Cmax was assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Pexidartinib
Number analyzed (Participants) | 7
ng/mL
  Pexidartinib | 12400 (32.2)
  ZAAD-1006a | 20400 (46.3)

10. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Participants Receiving Pexidartinib
Description: Tmax was calculated using standard non-compartmental analysis. Tmax for Pexidartinib and primary metabolite, ZAAD-1006a, are presented.
Time Frame: Week 3: Cycle 1 Day 1 at pre-dose, 0.5h, 1h, 2h, 4h, and 6h post-dose (each cycle is 28 days)
Population: Tmax was assessed in the Pharmacokinetic Analysis Set.
Measure: Median (Full Range); unit: hours
Arm/Group | Pexidartinib
Number analyzed (Participants) | 7
hours
  Pexidartinib | 2.08 [0.87 to 2.15]
  ZAAD-1006a | 2.12 [1.80 to 5.90]

ADVERSE EVENTS:
Time Frame: Adverse events (AE) were collected from the date of signing the informed consent form up post-treatment visit (28 ± 7 days after the last dose of study drug), up 13 months.
Description: A Treatment-emergent adverse event (TEAE) is defined as an AE that occurs, having been absent before the first dose of study drug, or has worsened in severity or seriousness after the initiating the study drug until post-treatment visit (28 ± 7 days after the last dose of study drug).
Arm/Group | Pexidartinib
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 6/40
Other Adverse Events (participants affected / at risk) | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pexidartinib (N=40)
Hepatic function abnormal (Hepatobiliary disorders) | 3
Fistula inflammation (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Epithelioid sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pexidartinib (N=40)
Hair color changes (Skin and subcutaneous tissue disorders) | 31
Pruritus (Skin and subcutaneous tissue disorders) | 19
Rash (Skin and subcutaneous tissue disorders) | 17
Skin discoloration (Skin and subcutaneous tissue disorders) | 7
Drug eruption (Skin and subcutaneous tissue disorders) | 5
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 5
Alopecia (Skin and subcutaneous tissue disorders) | 2
Urticaria (Skin and subcutaneous tissue disorders) | 2
Alanine aminotransferase increased (Investigations) | 24
Aspartate aminotransferase increased (Investigations) | 23
Blood lactate dehydrogenase increased (Investigations) | 19
Gamma-glutamyltransferase increased (Investigations) | 15
White blood cell count decreased (Investigations) | 14
Blood alkaline phosphatase increased (Investigations) | 12
Neutrophil count decreased (Investigations) | 11
Blood creatine phosphokinase increased (Investigations) | 8
Bilirubin conjugated increased (Investigations) | 6
Blood bilirubin increased (Investigations) | 6
Lymphocyte count decreased (Investigations) | 5
Blood cholinesterase increased (Investigations) | 3
Monocyte count decreased (Investigations) | 3
Blood cholesterol increased (Investigations) | 2
Blood triglycerides increased (Investigations) | 2
C-reactive protein increased (Investigations) | 2
High density lipoprotein increased (Investigations) | 2
Low density lipoprotein decreased (Investigations) | 2
Total bile acids increased (Investigations) | 2
Weight decreased (Investigations) | 2
Face oedema (General disorders) | 17
Fatigue (Investigations) | 12
Oedema peripheral (General disorders) | 4
Swelling face (General disorders) | 4
Asthenia (General disorders) | 2
Pyrexia (General disorders) | 2
Nausea (Gastrointestinal disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 5
Dry mouth (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 4
Abdominal distension (Gastrointestinal disorders) | 2
Gastrointestinal disorder (Gastrointestinal disorders) | 2
Dizziness (Nervous system disorders) | 4
Dysgeusia (Nervous system disorders) | 4
Headache (Nervous system disorders) | 3
Hypoaesthesia (Nervous system disorders) | 2
Memory impairment (Nervous system disorders) | 2
Taste disorder (Nervous system disorders) | 2
Periorbital oedema (Eye disorders) | 9
Eyelid oedema (Eye disorders) | 2
Decreased appetite (Metabolism and nutrition disorders) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 4
Hyperlipidaemia (Metabolism and nutrition disorders) | 3
Enzyme abnormality (Metabolism and nutrition disorders) | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 2
Anaemia (Blood and lymphatic system disorders) | 8
Leukopenia (Blood and lymphatic system disorders) | 3
Nasopharyngitis (Infections and infestations) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Hypertension (Vascular disorders) | 5
Hepatic function abnormal (Hepatobiliary disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-29): https://cdn.clinicaltrials.gov/large-docs/22/NCT04488822/Prot_SAP_000.pdf